CLINICAL TRIAL: NCT05693922
Title: Augmenting Single-session Behavioral Activation (BA) With Delta-beta Transcranial Alternating Current Stimulation (tACS) for the Treatment of Depression
Acronym: ABBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-2271
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
Keywords: transcranial alternating current stimulation; cross-frequency coupling; behavioral activation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants will take part in a single-session behavioral activation (BA) intervention. To examine the effects of neurostimulation on treatment response, participants will be randomized to receive either delta-beta cross-frequency transcranial alternating current stimulation (tACS) or an active sham.
Who Masked: Participant, Investigator
Masking Description: This study is designed to be double-blind. This means that the participant and the researchers are unaware of each participant's assignment until the completion of all data collection. This is accomplished using the randomization codes described above. Furthermore, this study utilizes an active sham stimulation. The active sham condition includes brief stimulation, mimicking the skin sensations associated with tACS. In our previously concluded trial, participants in the delta-beta tACS and active sham groups responded similarly to the blinding questionnaire, indicating that our active sham stimulation successfully blinded the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Delta-beta tACS (Experimental): Participants will receive a single session intervention of behavioral activation (BA) psychotherapy. Stimulation will be delivered via the NeuroConn DC-STIMULATOR MC at 1 milliampere (mA) zero-to-peak amplitude at the target electrodes and 2 mA zero to-peak amplitude at the return electrode. The tACS will be delivered using the cross-frequency stimulation waveform delta-beta (3-20Hz).
  Interventions: Device: Delta-beta cross-frequency transcranial alternating current stimulation via the NeuroConn DC-STIMULATOR MC; Behavioral: Single-session behavioral activation
- Active-sham tACS (Sham Comparator): Participants will receive a single session intervention of behavioral activation (BA) psychotherapy. The active sham condition includes brief stimulation, mimicking the skin sensations associated with tACS, assisting with blinding the participant's assignment.
  Interventions: Behavioral: Single-session behavioral activation; Device: Active sham cross-frequency transcranial alternating current stimulation via the NeuroConn DC-STIMULATOR MC

INTERVENTIONS:
Device: Delta-beta cross-frequency transcranial alternating current stimulation via the NeuroConn DC-STIMULATOR MC — Delta-beta stimulation will be delivered via the NeuroConn DC-STIMULATOR MC, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research.
  Arms: Delta-beta tACS
Behavioral: Single-session behavioral activation — Participants will take part in a single-session behavioral activation (BA) intervention. This intervention was adapted from standard BA protocols for the treatment of depression to be completed in a single, 90-minute session. This intervention will have 4 main components based on prior protocols:
  * Treatment overview and rationale
  * Tracking of daily activities
  * Exploration of values
  * Planning/scheduling activities
Device: Active sham cross-frequency transcranial alternating current stimulation via the NeuroConn DC-STIMULATOR MC — Active sham stimulation will be delivered via the NeuroConn DC-STIMULATOR MC, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research.
  Arms: Active-sham tACS

SUMMARY:
Investigating whether delta-beta cross-frequency transcranial alternating current stimulation can augment the effects of a single session of behavioral activation in participants with major depressive disorder.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether concurrent transcranial alternating current stimulation (tACS) augments the effects of a single session behavioral activation (BA) treatment of depression. Following a series of clinical assessments, participants will perform a reward-based decision-making task while electroencephalography (EEG) is collected.

Then, all participants will take part in a single-session 90-minute BA intervention; half of the participants will receive delta-beta tACS during the final 30 minutes of the session and half will receive an active sham stimulation. Participants will return two weeks later for another task-based EEG. Four weeks after the intervention session, they will receive self-report questionnaires via email to complete online.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or order
* Able to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Speak and understand English
* DSM-5 diagnosis of major depressive disorder (MDD) as assessed by the MINI

Exclusion Criteria:

* Participants must not have active suicide intent as determined by the Columbia Suicide Severity Rating Scale (C-SSRS). Active suicide intent will be captured in responses to items 4 and/or 5 on the C-SSRS.
* Participants must not meet criteria for current severe substance use disorder, anorexia nervosa, or active psychosis as captured by the MINI.
* Participants may not currently be in psychotherapy and have not received any other psychotherapy and/or stimulation (ECT, TMS) within the last 4 weeks.
* Any participants taking psychotropic medication must be on a stable dose for at least 4 weeks with no planned dose changes within the next 4 weeks.
* (for female participants) Participants must not be pregnant or breastfeeding.
* Participants may not have any medical or neurological illness for which symptom presentation or treatment could interfere with study participation
* Participants may not have undergone prior brain surgery
* Participants may not have any brain devices/implants, including cochlear implants and aneurysm clips
* Participants may not have had brain injury or concussion within the last three months
* Participants may not have a history of brain injury requiring current treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Delta-beta tACS: Participants will receive a 90- minute single session intervention of behavioral activation (BA) psychotherapy. Stimulation will be delivered during the final 30 minutes via the NeuroConn DC-STIMULATOR MC at 1 milliampere (mA) zero-to-peak amplitude at the target electrodes and 2 mA zero to-peak amplitude at the return electrode. The tACS will be delivered using the cross-frequency stimulation waveform delta-beta (3-20Hz).
  Delta-beta cross-frequency transcranial alternating current stimulation via the NeuroConn DC-STIMULATOR MC: Delta-beta stimulation will be delivered via the NeuroConn DC-STIMULATOR MC, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research.
- Active-sham tACS: Participants will receive a 90-minute single session intervention of behavioral activation (BA) psychotherapy. The active sham condition includes brief stimulation beginning in the final 30 minutes, mimicking the skin sensations associated with tACS, assisting with blinding the participant's assignment.
  Active sham cross-frequency transcranial alternating current stimulation via the NeuroConn DC-STIMULATOR MC: Active sham stimulation will be delivered via the NeuroConn DC-STIMULATOR MC, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research.
Period: Overall Study
Arm/Group | Delta-beta tACS | Active-sham tACS
Started | 15 | 15
Completed Week 2 Follow-Up | 15 | 12
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Delta-beta tACS: Participants will receive a 90- minute single session intervention of behavioral activation (BA) psychotherapy. Stimulation will be delivered during the final 30 minutes via the NeuroConn DC-STIMULATOR MC at 1 milliampere (mA) zero-to-peak amplitude at the target electrodes and 2 mA zero to-peak amplitude at the return electrode. The tACS will be delivered using the cross-frequency stimulation waveform delta-beta (3-20Hz).
- Active-sham tACS: Participants will receive a 90-minute single session intervention of behavioral activation (BA) psychotherapy. The active sham condition includes brief stimulation beginning in the final 30 minutes, mimicking the skin sensations associated with tACS, assisting with blinding the participant's assignment.
- Total: Total of all reporting groups
Arm/Group | Delta-beta tACS | Active-sham tACS | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (17.78) | 35.6 (13.56) | 36.2 (15.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 10 | 14 | 24
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinician-rated Depressive Symptoms
Description: Treatment response will be reported for clinician-rated depression symptom scores using the Hamilton Depression Rating Scale (HDRS). Items are scaled either from 0-2 to 0-4, and each item is summed for a total score ranging from 0 to 53 with higher scores indicating greater depression symptoms. Benchmarks suggested at: 0-7 normal; 8-13 mild depression; 14-18 moderate depression; 19-22 severe depression; >=23 very severe depression.
Time Frame: Baseline, 2 weeks post treatment
Population: Three participants randomized to the sham condition did not complete the follow-up visit. Missing data for these participants was handled using the intent-to-treat last value carried forward method.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delta-beta tACS | Active-sham tACS
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 19.33 (4.59) | 19.93 (4.71)
  2 weeks post treatment | 11.33 (5.15) | 13.93 (6.23)
Statistical Analysis 1: Comparison: Delta-beta tACS vs Active-sham tACS; Test type: Superiority; p = 0.34, ANOVA

2. Secondary Outcome: Phase-amplitude Coupling (PAC) Between Delta-beta Oscillations During Task Performance of the Streamlined Expenditure of Effort for Reward Task (S-EEfRT)
Description: Participants choose to complete a "hard" task or "easy" task. Coupling during the hard/easy decision is calculated between delta oscillations phase (2-3Hz) in prefrontal electrodes (FCz and surrounding electrodes) and the beta oscillations amplitude (15-25Hz) in left motor electrodes (C3 and surrounding electrodes). Instantaneous phase & amplitude of oscillations is calculated by averaging the signal in the two regions, band-filtering the signal to the specified range, and performing the Hilbert transform. PAC is normalized by creating a null distribution randomly shifting the beta time series by at least 10% of the number of time points. PAC is calculated between the delta-phase time series and each randomly shifted beta-amplitude time series. PAC is z-transformed relative to the null distribution. Values range from -3 to 3 and a score >=0.4 means the coupling is present. A higher value represents greater coupling strength which has been linked with greater cognitive processing.
Time Frame: Baseline, 2 weeks post treatment
Population: Data were not properly collected for some participants due to technical difficulties.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Delta-beta tACS | Active-sham tACS
Number analyzed (Participants) | 11 | 11
Z-score
  Baseline | 0.286 (0.606) | 0.290 (0.516)
  2 weeks post treatment | 0.286 (0.786) | 0.044 (0.655)
Statistical Analysis 1: Comparison: Delta-beta tACS vs Active-sham tACS; Test type: Superiority; p = 0.54, ANOVA

3. Secondary Outcome: Proportion of Hard Trials Chosen During the S-EEfRT
Description: In the Streamlined Expenditure of Effort for Reward Task (S-EEfRT), participants choose to complete a "hard" task requiring many button presses or an "easy" task with fewer button presses for variable monetary incentives. Number of button presses is individualized for each participant. Goal-directed behavior will be calculated as the proportion of "hard" tasks chosen across trials.
Time Frame: Baseline, 2 weeks post treatment
Population: Data were not properly collected for some participants due to technical difficulties.
Measure: Mean (Standard Deviation); unit: proportion of trials
Arm/Group | Delta-beta tACS | Active-sham tACS
Number analyzed (Participants) | 14 | 15
proportion of trials
  Baseline | 0.562 (0.158) | 0.521 (0.205)
  2 weeks post treatment: number analyzed (Participants) | 12 | 12
  2 weeks post treatment | 0.504 (0.188) | 0.454 (0.103)
Statistical Analysis 1: Comparison: Delta-beta tACS vs Active-sham tACS; Test type: Superiority; p = 0.865, ANOVA

4. Other Pre Specified Outcome: Change in Clinician-rated Anhedonia Symptoms Using SHAPS-C
Description: The Snaith-Hamilton Pleasure Scale-Clinician (SHAPS-C) is a clinician administered tool to assess symptoms of anhedonia. The SHAPS-C items use a Likert scale of 1-4, with higher scores reflecting greater pathology.
Time Frame: Baseline up to follow-up 2 weeks post treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through intervention visit (1 week later) and study follow-up visit (2 weeks after intervention), approximately 3 weeks total.
Arm/Group | Delta-beta tACS | Active-sham tACS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delta-beta tACS (N=15) | Active-sham tACS (N=15)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Tingling (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Warm Skin Sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Flickering Lights (Eye disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT05693922/Prot_SAP_000.pdf